CLINICAL TRIAL: NCT04872452
Title: Analysis of Cutaneous Nerve Biopsies in Gastrointestinal Motility Disorders
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigators departed institution prior to any recruitment
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB00146085
Record Dates: First submitted 2021-04-30; First posted 2021-05-04 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Small Fiber Neuropathy; Gastrointestinal Dysmotility
MeSH Terms: conditions — Small Fiber Neuropathy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Gastrointestinal dysmotility participants (Experimental)
  Interventions: Procedure: Skin biopsy
- Healthy participants (Other)
  Interventions: Procedure: Skin biopsy

INTERVENTIONS:
Procedure: Skin biopsy — Any combination of the following six 3-6mm skin biopsies may be taken: palm, dorsum of hand, calf, other non-genital and non-face (this last one includes areas for use as negative controls which are not on the distal limbs). No more than 6 biopsies will be taken at one time.The biopsy size 3-6mm and method (punch, shave or wedge) will be done depending on the biologic assay destined for the biopsy. While 3mm will be sufficient for microarray analysis, 6mm will be required for any cell sorting preceding microarray analysis.

SUMMARY:
This study is being done to evaluate cutaneous nerve biopsies from patients with refractory gastrointestinal motility disorders. The purpose of the study is to evaluate skin biopsies for signs of small fiber neuropathy in GI dysmotility patients, which may provide a better understanding of the underlying pathology of their condition. Specifically, identifying any small fiber neuropathy that may exist in the peripheral nervous system may help us to better understand the mechanism of presumed enteric neuropathy that may be involved in causing GI dysmotility.

DETAILED DESCRIPTION:
1. Gather basic, clinical information and perform small 3-6mm skin biopsies.
2. Identify characteristics of epidermal nerve fibers in patients with symptoms of gastrointestinal dysmotility
3. To isolate skin-derived precursor cells from skin biopsies and test their ability to generate neurons in vitro and in immune-deficient mouse models.

ELIGIBILITY:
Inclusion Criteria:

* Individual with a gastrointestinal motility disorder that has failed both clinical and surgical options for symptomatic management

Exclusion Criteria:

* Child 17 years of age or younger
* Individuals incapable of informed consent
* Patient with diseased skin or on drugs which affect skin biology.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-12-22 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Presence of small fiber neuropathy in skin biopsy samples | Only one biopsy but analysis may take one year.
  Presence or absence of small fiber neuropathy obtained after the skin biopsy procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Pankaj J Pasricha, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States